CLINICAL TRIAL: NCT06052371
Title: VerioVue Enhancements Regulatory Clinical Evaluation - Professional Comparison to Validated Method: Neonate Study
Brief Title: Project VerioVue Enhancements - Neonate Study
Status: Terminated | Type: Observational
Why Stopped: This study was terminated for business reasons.
Sponsor: LifeScan Scotland Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: FILE-PROT-005443
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
Keywords: Neonate
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates: Newborn babies who are 28 days old or less with a corrected gestational age of at least 34 weeks and a weight of at least 1700g or more at the time of participation. They will be recruited from hospital neonatal units or wards.
  Interventions: Device: VerioVue (Enhancements) blood glucose monitoring system

INTERVENTIONS:
Device: VerioVue (Enhancements) blood glucose monitoring system — VerioVue meter with expanded haematocrit range
  Other Names: OneTouch VerioVue blood glucose monitoring system

SUMMARY:
The goal of this performance evaluation is to compare the blood glucose results obtained using the VerioVue Blood Glucose Monitoring system (BGMS) with those obtained from a validated comparator method (iSTAT 1 Analyser) using blood obtained from neonates. The main question it aims to answer is:

•How accurate is the VerioVue BGMS when compared to a product that has already been confirmed as accurate (iSTAT 1 Analyser) when hospital staff test blood taken from neonates on these instruments? Participants (neonates) will have a small amount of blood taken from a heel prick (performed by a HCP for medical purposes) or from an existing arterial line.

DETAILED DESCRIPTION:
UK NHS Hospital sites (between 1 and 3 sites) will be used to collect a minimum of 200 evaluable blood samples from neonates meeting the inclusion criteria. Consent will be taken from the neonates parent prior to participation in the study. They will consent to one or two blood samples to be taken from their child. If the participant meets the enrolment criteria then demographics and prescription medication (including dietary supplements) information will be collected. A small volume of blood (max 150µl) will be collected from an existing arterial line or from a heel prick that is being performed for medical purposes. This blood will then be applied to six investigational One Touch VerioVue meters (with expanded haematocrit range of 20-65%) fitted with OneTouch Verio test strips and the blood glucose meter readings recorded. Three different lots of test strips will used in rotation across the study. Within 5 minutes of the last meter test, NHS study staff will use blood from the same sample and perform a test on the iSTAT 1 Analyser to obtain blood glucose, haematocrit and oxygen levels of the sample. No treatment decisions will be made based on the blood glucose results obtained for this study. The study documentation will be reviewed by LifeScan monitors for completeness and accuracy and the results entered into a validated database. The data will be extracted and statistically analysed to determine the accuracy of the blood glucose results obtained using the OneTouch VerioVue BGMS when compared to the blood glucose results obtained on the iSTAT 1 Analyser.

ELIGIBILITY:
Inclusion Criteria:

* Age - Newborn babies, 28 days old or less with a corrected gestational age of at least 34 weeks and a weight of at least 1700g or more at the time of participation.
* Informed Consent - Study participants parents must read the Parental Participant Information Sheet and sign the Parental Informed Consent Form
* Study participants parent agrees to provide information related to demographics, prescription medication, dietary supplements, and results from other physician ordered testing e.g., Bilirubin (total, conjugated, and unconjugated) where available.
* Study participants parent agrees to allow study staff access to medical records where necessary.
* Study participants parents agree to all aspects of the study process, including where applicable arterial blood draw from an existing arterial line or a heel prick performed by an HCP for medical purposes.

Exclusion Criteria:

* Age- Newborn more than 28 days old.
* Study participants with a gestational age of less than 34 weeks at the time of participation.
* Study participants with a gestational weight of less than 1700g
* Current positive test result for Covid-19.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates will be enrolled into the study from NHS hospital neonatal units and wards.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Performance evaluation: blood glucose monitoring system accuracy: BGMS vs reference instrument | 1 hour
  Performance Evaluation to compare the VerioVue BGMS blood glucose results to results obtained using the iSTAT 1 Analyser, a validated comparator method.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Zammitt, MBCHB, Principal Investigator — Edinburgh Centre for Endocrinology and Diabetes
Locations (3):
- United Kingdom (3):
  - Whipps Cross University Hospital (Barts Health NHS Trust), London
  - Queens Hospital Romford (BHRUT), London
  - The Royal Oldham Hospital (Northern Care Alliance NHS Foundation Trust), Manchester

IPD SHARING:
Plan to Share IPD: No